CLINICAL TRIAL: NCT02637466
Title: A Double-blind, Placebo-controlled, Randomized Study of Vortioxetine Treatment on Major Depression, Cognition, and Systemic Inflammatory Biomarkers Associated With Depression and Cancer Progression in Women With Breast Cancer.
Brief Title: Vortioxetine for MDD, Cognition, and Systemic Inflammatory Biomarkers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not received
Sponsor: University of Miami (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Dominique Musselman, Principal Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150753
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Unipolar Major Depression; Stage I, II or III Breast Cancer
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vortioxetine (Experimental): In cycle I of the study, participants will be randomized on to flexible-dose VTX (10-20 mg) versus. Vortioxetine starting dose will be 10 mg daily. Vortioxetine starting dose will be 10 mg daily with a dose escalation up to 20 mg daily at week #4. Study cycle II is an 8-week, open label treatment design for non-responders completing the Cycle I RCT. One treatment arm will continue VTX non-responders to 8 week VTX (10-20 mg/day) augmentation with cognitive behavioral therapy (10 sessions). The 2nd treatment arm will continue placebo non-responders who complete the RCT to VTX (10 to 20 mg/day). The third treatment arm will continue VTX responders/remitters who complete the RCT to open-label VTX for another 8-weeks to assess maintenance efficacy for up to 16 weeks.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): In cycle I of the study, 80 eligible depressed women with breast cancer will be randomized into an 8-week, double-blind, placebo-controlled, flexible-dose vortioxetine (10-20 mg) treatment arm versus placebo arm.
  Responders to placebo treatment will complete their study participation at the end of Cycle I, and will not proceed to Cycle II.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine
  Other Names: Brilliantex

SUMMARY:
The purpose of this antidepressant study is to determine the efficacy of vortioxetine on depression and cognition in 80 women with breast cancer, and to elucidate inflammatory-mediated mechanisms by which depression and its treatment influence cancer outcome. Our hypothesis is that effective vortioxetine antidepressant therapy in depressed women with breast cancer will attenuate increased intermediate endpoints of inflammation that contribute to the pathogenesis of depression, cognitive impairment, and cancer progression

DETAILED DESCRIPTION:
Major depression is an independent risk factor for incident cancer, recurrence and mortality. Women with chronic major depression exhibit a four-fold increased rate of incident breast cancer and a 39% higher mortality rate compared to non-depressed women with breast cancer. Although the precise biological mechanism linking depression with cancer progression remains unclear, elevated concentrations of systemic inflammatory biomarkers (e.g., pro-inflammatory cytokine interleukin-6 (IL-6) and associated cytokine proteins) have been independently associated with depression and cancer progression. In the context of breast cancer, secretion of tumor-derived cytokines is a known mechanism by which epithelial tumors are able to recruit immune cells (MDSCs). The presence of MDSCs at the primary tumor site favors tumor pathogenesis and correlates with more aggressive breast cancer subtypes. At the systemic level, increased levels of interleukin-6, circulating MDSCs, circulating tumor cells (CTCs) and inflammatory markers in the bloodstream of breast cancer patients are found to strongly correlate with poor prognosis.

Medical conditions such as major depression are associated with increased levels of systemic pro-inflammatory cytokines, thereby creating a host environment that promotes cancer progression. Indeed, innate immune activation and chronic inflammation have been implicated in the pathogenesis of major depression and may account for the biological mechanism linking depression and cancer progression. Several studies have shown antidepressant treatment response attenuates and normalizes pro-inflammatory cytokine plasma levels in medically-healthy patients with depression. To date, only three randomized controlled antidepressant studies have been conducted in depressed women with breast cancer. Two studies found mainserin to be effective and superior to placebo, whereas paroxetine and desipramine were comparable to placebo. Notably, several randomized controlled trials in depressed breast cancer patients found psychotherapy to be an effective depression treatment. Moreover, these studies found psychotherapy significantly lengthened survival time in depressed breast cancer patients with metastatic disease. Remarkably, no randomized controlled trials have examined the impact of antidepressant medications on cancer survival.

To date, there have been no randomized, placebo-controlled antidepressant studies in depressed women with breast cancer to investigate the impact of depression treatment on cognition and the inflammatory mediators that promote cancer progression. This study will explore the efficacy of vortioxetine on depression and cognition in women with breast cancer, and determine whether successful treatment of depression alters circulating cytokines, immune mediators, and circulating tumor cells, thus elucidating a possible mechanism to explain improved cancer outcome with effective antidepressant treatment. Given the disproportionately high rate of depression in women with breast cancer and its negative impact on cancer outcome, understanding the biological mechanism that drives this relationship is critical. This study may uncover novel immune-mediated mechanisms by which vortioxetine treatment ameliorates depression, enhances cognition, and influences cancer outcome.

Primary Objective - To assess antidepressant efficacy of vortioxetine (VTX) treatment in women with major depressive disorder (MDD) who have completed curative treatment of Stage I, II or III breast cancer.

Primary Endpoint Antidepressant efficacy will be assessed by the Hamilton Depression Rating Scale-21 (HDRS-21) total score administered at specified time points. Antidepressant response is defined as a 50% reduction in baseline HDRS-21 total score, and treatment remission is defined as an HDRS-21 total score ≤7. Antidepressants will be deemed effective if the patient's depression does not worsen. A participant's depression will be classified as "worse" if a) the participant becomes suicidal or psychotic, b) their HAM-D score increases > 18, or over a four-week period of time: c) the HAM-D score increases, and d) the CGI Improvement Rating has increased by at least one point. The definitions of antidepressant efficacy and worsening depression remain the same during Cycle 2.

- Cognitive function will be assessed by Brief Assessment of Cognition in Affective Disorders (BAC-A) test battery with measures in: (1) list learning, (2) digit sequencing task, (3) token motor task, (4) verbal fluency, (5) tower of London test, (6) symbol coding, and (7) affective processing subtest. All BAC-A measures will be administered at specified time points, and the total composite z-scores will be compared to baseline total composite z-scores.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 to 75 years of age
2. Confirmed diagnosis of Stage I, II, or III breast cancer
3. Completed curative cancer treatment (surgery, chemotherapy, and/or radiotherapy) at least four weeks (≥ 4 weeks) prior to study entry no more than 5 years.
4. Unipolar major depression confirmed by the mood disorder module in Structured Clinical interview for DSM-V (SCID)
5. Baseline depression severity total score ≥18 by Hamilton Depression Rating Scale-21 (HDRS-21)
6. Negative urine pregnancy test in women of child-bearing potential (WOCBP).
7. Use of medically-established contraceptive method (e.g., contraceptive hormone therapy or intrauterine device) in women of child-bearing potential (WOCBP) or abstinence from heterosexual intercourse from the time of signing informed consent through 14 days after the last dose of study drug.
8. Ability to understand and the willingness to sign a written informed consent and HIPAA document/s

Exclusion Criteria:

* 1. Other active cancers [EXCEPTION: cured skin cancer]. 2. Actively suicidal, as determined by certified mental health provider. 3. Comorbid bipolar disorder or psychosis, as diagnosed by psychiatric clinical interview conducted by a certified mental health provider.

  4. Mini-mental state exam (MMSE) score <24 at baseline assessment 5. Current use of stimulant and/or amphetamine for cancer-related fatigue or cognitive impairment.

  6. Use of current and effective antidepressants during study period. [NOTE: Patients who have not responded to current antidepressant may be tapered off medication prior to study entry.] 7. Uncontrolled hypothyroidism. Must be biochemically (TSH, T3, T4) and clinically euthyroid at baseline assessment.

  8. Use of monoamine oxidase inhibitors (MAOIs) in past 14 days. 9. Concomitant use of mood stabilizer including lithium, lamictal and atypical antipsychotics 10. Failed prior therapy with vortioxetine (VTX) 11. Positive urine toxicology screen for cocaine, opiates, marijuana, amphetamines.

  12. Comorbid alcohol and/or substance use disorder within the prior 12 months of screening, as diagnosed by psychiatric clinical interview conducted by a certified mental health provider.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Antidepressant efficacy | 4-16 weeks
  Antidepressant efficacy will be assessed by the Hamilton Depression Rating Scale-21 (HDRS-21) total score administered at specified time points. Antidepressant response is defined as a 50% reduction in baseline HDRS-21 total score, and treatment remission is defined as an HDRS-21 total score ≤7. Antidepressants will be deemed effective if the patient's depression does not worsen. A participant's depression will be classified as "worse" if a) the participant becomes suicidal or psychotic, b) their HAM-D score increases > 18, or over a four-week period of time: c) the HAM-D score increases, and d) the CGI Improvement Rating has increased by at least one point. The definitions of antidepressant efficacy and worsening depression remain the same during Cycle 2.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Musselman, M.D., MSCR, Principal Investigator — University of Miami